CLINICAL TRIAL: NCT03439826
Title: Junior / Senior Concordance in Ultrasound Assessment of Crohn's Disease (ECHOCROHN)
Brief Title: Junior / Senior Concordance in Ultrasound Assessment of Crohn's Disease
Acronym: ECHOCROHN
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3094_ECHOCROHN
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory disease of the intestine (IBD), evolving with varying periods of remissions and relapses, characterized by segmental inflammation of the digestive tract, which can be complicated by stenosis, fistulas or even digestive cancers.

The emergence of effective therapeutic strategies has led to the adoption of more ambitious therapeutic objectives that have no longer the improvement of symptoms but a complete cicatrization of the intestinal mucosa as an objective.

The disadvantage of the latter is the need for its evaluation by ilo-colonoscopy, "gold-standard", invasive, not without risks (perforation, anesthesia, hemorrhage), requiring colonic preparation and hospitalization.

In this context, the use of non-invasive markers performed in routine practice (hemogram, VS, CRP, fibrinogen, fecal calprotectin, abdominal ultrasound), predictive of this endoscopic mucosal healing, is a necessity to improve the tolerance of follow-up and allow better adherence by the patient of the therapeutic project. A decrease in health costs could also be associated with the use of these markers.

Abdominal ultrasound is an accessible, inexpensive, non-invasive and non-irradiating imaging medium. It is very useful and has proved its effectiveness in monitoring Crohn's disease to evaluate the activity of the disease in order to predict mucosal healing and to detect complications (stenosis, fistula, abscess) (1, 2, 3). However, especially for the study of the small intestine this act is known to be very dependent on the operator and the conditions of examination (echogenicity of the patient). In addition, few objective criteria have been described in the literature for the study of Crohn's disease (2, 3).

A recent study under submission has developed an ultrasound score of Crohn's disease activity, which through the study of each segment (distal ileum, right colon / transverse / left, sigmoid) using 14 criteria , allowed to rule on the activity of the disease and thus to predict mucosal healing. In this study, which concerned 48 patients, ultrasound scans were performed by radiologists experienced in abdominal pathology. This score was very easy to use and powerful to study the disease activity of each segment with 2 parameters in particular: parietal thickness and changes in fat.

It therefore seems necessary to confirm the simplicity of this ultrasound score in a validation cohort to: in particular to study the inter-observer reproducibility so as to be able to extend the use of this score to non-specialist radiologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed for Crohn's disease;
* Crohn's disease diagnosed in accordance with the criteria of the European Crohn's and Colitis Organization (ECCO);
* Benefiting from an abdominal ultrasound as part of their usual follow-up;
* Not having expressed his opposition to participate in the study.

Exclusion Criteria:

* Persons of legal age subject to legal protection (protection of justice, guardianship, tutorship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Inter-observer reproducibility (junior / senior) of an ultrasound score of Crohn's disease activity | Baseline
  These criteria are to be found on each segment: terminal ileum, right colon, transverse colon, left colon and sigmoid.
  * Normal appearance: yes / no
  * Maximum parietal wall thickness (mm)
  * parietal differentiation: yes / no
  * Ulceration: yes / no
  * Fistula: yes / no
  * Infiltration of peripheral fat: yes / no
  * Sclerolipomatosis: yes / no
  * Stenosis: yes / no
  Criterion for the entire abdominal cavity :
  * Mesangular ganglion> 5mm: yes / no
  * Intraperitoneal fluid effusion: yes / no Abdominal abscess: yes / no
  * dilated handles: yes / no
  * Total length of reach (in mm)
  * Distance to the valve

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Bouguen, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France